CLINICAL TRIAL: NCT00986882
Title: A Double-blind, Randomized, Single Dose, Placebo Controlled, Three Part Study to Evaluate the Safety and Tolerability, Efficacy and Dose Response of SAF312 in Postoperative Dental Pain Patients
Brief Title: To Evaluate the Safety, Tolerability and Analgesic Efficacy of SAF312 in Postoperative Dental Pain Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSAF312A2103
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-09

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAF312A (2 doses in part B; 5 - 6 doses in part C) (Experimental)
  Interventions: Drug: SAF312A
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Ibuprofen (Active Comparator)
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: SAF312A
  Arms: SAF312A (2 doses in part B; 5 - 6 doses in part C)
Drug: Placebo
  Arms: Placebo
Drug: Ibuprofen
  Arms: Ibuprofen

SUMMARY:
The study will assess the analgesic efficacy and safety and tolerability of a single oral dose of SAF312 in postoperative dental pain patients after 3rd molar extraction.

ELIGIBILITY:
Inclusion Criteria:

* Extraction of two or more impacted (partial or full) third molars. At least one of the impaction should be lower jaw.
* Each patient will evaluate her/his post-surgical pain intensity prior to taking trial medication.
* To be eligible for this trial, post surgical pain must be moderate to severe -- Subjects should be in good health otherwise as determined by past medical history, physical examination, vital signs, electrocardiogram and laboratory tests at screening.
* Female subjects should be either postmenopausal or should have had surgical sterilization.

Exclusion Criteria:

* Patients with known hypersensitivity to diclofenac, aspirin, acetaminophen or to antipyretics or with allergies manifested by attacks of asthma, urticaria or acute rhinitis following treatment with aspirin or other agents with cyclooxygenase-inhibiting activity such as NSAIDs.
* Use of antipyretic/analgesic drugs from 48 hrs pre-dose to 24 hrs postdose
* Presence of bleeding disorder (history of excessive bleeding after dental procedures or minor injuries)
* Patients with Diabetes mellitus.
* Presence, history of, or family history of malignant hyperthermia or anesthesia-related events that may be suggestive of malignant hyperthermia.
* An abnormal ECG at screening, including PR>200 ms, QRS>110 ms, QTcF<380 or >450 ms, lead II T wave abnormalities. Non-specific T wave abnormalities in leads other than lead II are permissible if not accompanied by any other morphological abnormalities.
* Patients with infection e.g. dental abscess

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 183 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety, tolerability, efficacy and dose response of single oral doses of SAF312 in patients with postoperative dental pain | 24 hours

SECONDARY OUTCOMES:
To assess the pharmacokinetics of the single oral doses of SAF312 and Ibuprofen in patients with postoperative dental pain | 24 hours
To measure: time-specific pain relief (PR), Total pain relief (TOTPAR), time to onset of analgesia, time to rescue medication | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mangwani-Mordani S, Goodman CF, Galor A. Novel Treatments for Chronic Ocular Surface Pain. Cornea. 2023 Mar 1;42(3):261-271. doi: 10.1097/ICO.0000000000003193. Epub 2022 Dec 19. PMID 36729473
- See also: Results for CSAF312A2103 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=6323